CLINICAL TRIAL: NCT02657018
Title: Mobile Exergaming for Health - Effects of a Serious Game Application for Smartphones on Physical Activity and Exercise Adherence in Type 2 Diabetes Mellitus (Randomized Controlled Trial)
Brief Title: Mobile Exergaming in Type 2 Diabetes
Acronym: MOBIGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Prof. Arno Schmidt-Trucksäss MD, MA, FESC, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EKNZ 2015-424
Record Dates: First submitted 2016-01-11; First posted 2016-01-15 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Overweight; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): MOBIGAME group
  Interventions: Device: MOBIGAME
- Control (Active Comparator): Lifestyle counseling group
  Interventions: Other: Control

INTERVENTIONS:
Device: MOBIGAME — Mobile phone based game-like software application and platform (MOBIGAME) that includes individualized and structured exercise regimens (endurance, strength, balance and flexibility) that are based on the user's individual fitness evaluation (through established fitness tests) and incorporated into the story line of a gardening simulation game.
  Arms: Intervention
Other: Control — One-time standard lifestyle counseling including the promotion of baseline activities of daily life as well as a structured exercise plan including strength and endurance exercises with moderately increasing intensity and duration that is to be implemented autonomously.
  Arms: Control

SUMMARY:
The purpose of this study is to investigate if MOBIGAME (an innovative, mobile phone-based game application) is suitable to increase daily physical activity and physical activity adherence as well as health parameters such as cardiorespiratory fitness, leg strength, glucose metabolism, vascular health and self-determination as well as health related quality of life in the course of a 24-week intervention in comparison to the control group receiving one-time lifestyle counseling.

DETAILED DESCRIPTION:
In recent years, type 2 diabetes mellitus (T2DM) has grown into an emerging pandemic that is a key determinant of morbidity and mortality in both developed and developing countries worldwide. The successful treatment and prevention of T2DM is one of the biggest future health care challenges and most important to manage the enormous socio-economic burden that is associated with T2DM and its various comorbidities. Physical inactivity is known to be one of the most important risk factors for the development of obesity and T2DM. In contrast, increases in physical activity (PA) and fitness can lower the T2DM incidence, improve the patient's glucose metabolism and reduce morbidity and (premature) mortality, independent of body mass index (BMI) or other risk factors. Despite the obvious benefits of regular PA in the treatment and prevention of T2DM, most activity-promoting programs targeting T2DM patients are seldom successful in the long term due to diminishing patient motivation. A novel approach to motivate those individuals that are the least likely to engage in regular PA to be more physically active and adhere to regular PA are active video games or "exergames" that combine PA and video gaming. However, existing exergames do not offer fitness-level adjusted, individualized workouts and are normally stationary and bound to a TV, thus not enabling PA anywhere and at any time. To address these shortcomings, the investigators used sports scientific expertise to develop a smartphone-based, mobile gardening simulation game application, specifically designed for middle-aged T2DM patients, to induce a healthier, more active lifestyle as part of a successful T2DM treatment and management.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Non-insulin-dependent diabetes mellitus (doctor diagnosed)
* Body Mass Index >25 kg/m2
* Regular smartphone use during the last year before the study
* Motivation to participate in the study for its entire duration of 24 weeks

Exclusion Criteria:

* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Previous enrolment into the current study
* Participation in other studies in the last four weeks
* Systolic blood pressure > 170mmHg, diastolic blood pressure > 100 mmHg
* Regular physical activity before the study (≥150 min moderate intensity daily PA per week or >1 endurance or strength training session per week of more than 30 min in duration)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline daily physical activity at 24 weeks | Baseline and 24 weeks
  Measured as steps per day.

SECONDARY OUTCOMES:
Adherence to the intervention | 24 weeks
  Measured as usage log entries (intervention group) and self-reported exercise log entries (control group).

OTHER OUTCOMES:
Change from baseline self-determination at 24 weeks | Baseline and 24 weeks
  Self-determination (intrinsic motivation, perceived competence, perceived choice, perceived usefulness measured via the score in an abridged, 12-item version of the Intrinsic Motivation Inventory.
Change from baseline cardiorespiratory fitness at 24 weeks | Baseline and 24 weeks
  Aerobic capacity measured as VO2peak.
Change from baseline six minute walking distance at 24 weeks | Baseline and 24 weeks
  Measured via the Six Minute Walk Test
Change from baseline isometric leg strength at 24 weeks | Baseline and 24 weeks
  Measured as maximal isometric force and rate of force development.
Change from baseline leg strength endurance at 24 weeks | Baseline and 24 weeks
  Assessed as maximum number of repetitions in the Sit-to-Stand Test (STS)
Change from baseline glucose metabolism at 24 weeks | Baseline and 24 weeks
  Fasting glucose, glycated hemoglobin (HbA1c), fasting C-peptides, fasting insulin levels and insulin resistance, measured as homeostasis model assessment (HOMA) index.
Change from baseline inflammatory markers at 24 weeks | Baseline and 24 weeks
  Total cholesterol, LDL- and HDL-cholesterol, triglycerides, apolipoprotein B, irisin, adiponectin and interleukin-6
Change from baseline central blood pressure at 24 weeks | Baseline and 24 weeks
Change from baseline pulse wave reflection at 24 weeks | Baseline and 24 weeks
  Measured as augmentation index.
Change from baseline arterial stiffness at 24 weeks | Baseline and 24 weeks
  Measured as aortic pulse wave velocity.
Change from baseline microvascular function at 24 weeks | Baseline and 24 weeks
  Measured as retinal vessel diameters.
Change from baseline health-related quality of life (HRQOL) at 24 weeks | Baseline and 24 weeks
  Assessed with score in the 36-item Short Form questionnaire (SF-36).
Change from baseline fatigue at 24 weeks | Baseline and 24 weeks
  Measured via the score in the 13-item FACIT Fatigue Scale.
Perceived acceptance of intervention | 24 weeks
  Measured via the Technology Acceptance Model (TAM) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, MD, MA, FESC, Principal Investigator — University of Basel
Locations (1):
- Division of Sports and Exercise Medicine, Department of Sport, Exercise and Health, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hochsmann C, Muller O, Ambuhl M, Klenk C, Konigstein K, Infanger D, Walz SP, Schmidt-Trucksass A. Novel Smartphone Game Improves Physical Activity Behavior in Type 2 Diabetes. Am J Prev Med. 2019 Jul;57(1):41-50. doi: 10.1016/j.amepre.2019.02.017. Epub 2019 May 22. PMID 31128953
- [Derived] Hochsmann C, Infanger D, Klenk C, Konigstein K, Walz SP, Schmidt-Trucksass A. Effectiveness of a Behavior Change Technique-Based Smartphone Game to Improve Intrinsic Motivation and Physical Activity Adherence in Patients With Type 2 Diabetes: Randomized Controlled Trial. JMIR Serious Games. 2019 Feb 13;7(1):e11444. doi: 10.2196/11444. PMID 30758293
- [Derived] Hochsmann C, Walz SP, Schafer J, Holopainen J, Hanssen H, Schmidt-Trucksass A. Mobile Exergaming for Health-Effects of a serious game application for smartphones on physical activity and exercise adherence in type 2 diabetes mellitus-study protocol for a randomized controlled trial. Trials. 2017 Mar 6;18(1):103. doi: 10.1186/s13063-017-1853-3. PMID 28264717